CLINICAL TRIAL: NCT02694562
Title: Microparticle Enhanced Cytotoxic Transarterial Embolization Therapy: A Pilot Study of Irinotecan in the Treatment of Metastatic Colorectal Carcinoma (mCRC) by Embozene TANDEM™ Drug-Eluting Microspheres Embolization
Brief Title: Microparticle Enhanced Cytotoxic Transarterial Embolization Therapy
Acronym: MIRACLEIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRACLE III
Record Dates: First submitted 2016-02-25; First posted 2016-02-29 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Carcinoma
Keywords: Metastatic Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 40um Embozene TANDEM Microspheres (Experimental): 40um Embozene TANDEM Microspheres loaded with Irinotecan (up to 150 mg)
  Interventions: Device: 40um Embozene TANDEM Microspheres

INTERVENTIONS:
Device: 40um Embozene TANDEM Microspheres — 40um Embozene TANDEM Microspheres loaded with Irinotecan (up to 150 mg).

SUMMARY:
The purpose of this study is to determine safety and local tumor control of Embozene TANDEM Microspheres (40um TANDEM) loaded with Irinotecan to treat metastatic colorectal carcinoma (mCRC).

DETAILED DESCRIPTION:
Colon or rectal carcinoma that has spread to the liver is considered to be metastatic and is a Stage IV cancer. If the metastasized tumor is unresectable, the only current treatment is chemotherapy. Transarterial Chemoembolization (TACE) is considered as a palliative treatment in advanced metastatic colorectal carcinoma (mCRC), with the potential of local tumor control. TACE has evolved in the past 8 years to include drug-delivery devices that can target and deliver drugs from small microparticles (DEB-TACE). Superselective DEB-TACE has the potential to penetrate deeper into the tumor's vasculature to reach peripheral growing points. Loading these microparticles with a cytotoxic drug may improve the level of local tumor control.

The MIRACLE III study is a controlled, pilot, single center (Italy) study on 18 subjects with pretreated non-resectable mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age >18 yrs who have histologically confirmed adenocarcinoma of the colon or rectum (Stage IV)
* Presence of metastatic disease with liver as dominant disease-site defined as >80% tumor body burden confined to liver; less than 60% liver tumor replacement.
* Subject is competent and willing to provide written informed consent in order to participate in the study.
* Eastern Cooperative Oncology Group (ECOG) performance status is 0-1 or Child-Pugh classification is A or B7.
* Multinodular or single nodular tumor 4 cm, patients with bilobar disease who can be treated superselectively in a single session or both lobes able to be treated within 3 weeks. Patient must have at least one tumor lesion that meets the following criteria: lesion can be accurately measured in at least one dimension according to the Modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.
* Pretreatment with two or more lines of chemotherapy containing Fluorouracil (5-FU) or analogue, oxaliplatin, irinotecan ± bevacizumab ±epidermal growth factor receptor (EGFR)-inhibitors, if indicated, for metastatic disease.
* No invasion in the blood vessel (hepatic portal, hepatic vein) or bile duct by the computerized axial tomography (CT) or Magnetic Resonance (MR) Imaging.
* Proper blood, liver, renal, heart function: testing result within 2 weeks from registry of this study as follows:

  1. White Blood Cell (WBC) >3,000 cells/mm3
  2. Absolute neutrophil count ≥1500/mm3
  3. International Normalized Ratio (INR) <2.0
  4. Partial Thromboplastin Time (PTT) <40 sec
  5. Platelet count >50,000/mm3
  6. Blood bilirubin <3.0 mg/dL
  7. Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT) is within 5 times of normal range of each organ
  8. Serum creatinine <1.5 mg/dL
  9. Hemoglobin >8.0 g/dL
  10. Alkaline phosphatase <630 IU/L
  11. No unstable coronary artery disease or recent Myocardial Infarction(MI)
  12. Normal electrocardiogram (ECG) with QT interval <480 msec within the previous 12 months
  13. No current infections requiring antibiotic therapy
  14. Not on anticoagulation or suffering from a known bleeding disorder.
* Measureable disease per mRECIST.
* Expected survival more than 3 months

Exclusion Criteria:

* ECOG performance status >2; or Child-Pugh class>11 points or more, or American Society of Anaesthesiologists' (ASA) class 5 .
* Bilirubin levels >3 mg/dL
* mCRC within the large vessel or biliary duct invasion, diffuse hepatocellular carcinoma (HCC) or extrahepatic spread.
* Patients in which any of the following are contraindicated or present:

  1. The use of irinotecan
  2. MRI or CT scans
  3. Hepatic embolization procedures
  4. WBC <3000 cells/mm3
  5. neutrophil <1500 cells/mm3
  6. Cardiac ejection fraction <50% assessed by isotopic ventriculography, echocardiography or MRI
  7. Elevated serum creatinine ≥ 2.5 mg/dL
  8. Impaired clotting test (platelet count < 50,000/mm3, PT-INR >2.0
  9. AST and/or ALT >5x upper limit of normal (ULN), when greater >250 U/I
  10. Known hepatofugal blood flow.
  11. Arterio-venous shunt
  12. Arterio-portal shunt
  13. Main stem portal vein occlusion
* Women who are pregnant or nursing
* Allergy to iodinated contrast used for angiography
* Tumour burden of more than 50% of liver volume (Tumor volume by be smaller e.g. ≤30%)
* Patients with active bacterial, viral (HIV), or fungal infection.
* Other malignancies
* Any co-morbid disease or condition or event that, in the investigator's judgment, would place the patient a undue risk what would preclude the safe use of DEB-TACE.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Orsi, MD, Principal Investigator — European Institute of Oncology (Milan Italy)
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty MIRACLE III subjects were consented. Of these 20, eighteen (18) were enrolled and treated in the trial. Two subjects were not enrolled as they did not meet I/E criteria. These two subjects have been reported as screen failures.
Period: Overall Study
Arm/Group | 40um Embozene TANDEM Microspheres
Started | 20
Completed | 2
Not Completed | 18
Not completed — Death | 8
Not completed — Protocol Violation | 4
Not completed — Lost to Follow-up | 3
Not completed — Screen Failure | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: A total of 20 patients were consented to participate however, 2 patients were not enrolled as they were reported as screen failures prior to the first study treatment. Therefore a total of 18 baseline patients were assessed.
Arm/Group | 40um Embozene TANDEM Microspheres
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 18
Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — ECOG 0 - Fully active, able to carry out all pre-disease performance without restriction. ECOG 1 - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work. ECOG 2 - Ambulatory and capable of all self care, but unable to carry out any work activities. Up and about more than 50% of waking hours. ECOG 3 - Capable of only limited self care, confined to bed or chair more than 50% of waking hours. ECOG 4 - Completed disabled. Cannot carry out any self care. Totally confined to bed or chair. ECOG 5 -Dead
  Participants
    ECOG Score 0 | 18
    ECOG Score 1 | 0
    ECOG Score 2 | 0
Classification of Malignant Tumours (TNM) Stage [Count of Participants; unit: Participants] — TNM staging takes into account the size of the tumour, whether the lymph nodes (glands) are affected and whether cancer cells have spread anywhere else.
  TNM stands for Tumour, Node, Metastasis. The TNM system describes the size of a primary tumour (T), whether the cancer has spread to the lymph nodes (N), and whether the cancer has spread to a different part of the body (M - for metastases).
  Participants
    TNM Stage I | 0
    TNM Stage II | 0
    TNM Stage III | 0
    TNM Stage IV | 18
Child Pugh [Count of Participants; unit: Participants] — The Pugh-Child score is measured utilizing five clinical measures. The five measures are: total bilirubin (yellow compound in bile from hemoglobin breakdown), serum albumin (blood protein produced in the liver), prothrombin time (time for blood to clot), ascites (fluid in peritoneal cavity), and hepatic encephalopathy (brain disorder from liver disease). A score of 1, 2, or 3 is given to each measure, with 3 being the most severe.
  From these assessments, Child-Pugh is scored as follows: Class A (5 to 6 points), Class B (7 to 9 points), and Class C (10 to 15 points)
  Participants
    Child Pugh - A | 17
    Child Pugh - B7 | 0
    Not Available | 1
History of Radiotherapy [Count of Participants; unit: Participants] | 2
History of Surgical Therapy [Count of Participants; unit: Participants] | 16
History of Systemic Therapy [Count of Participants; unit: Participants] | 18
Previous Lines of Chemotherapy [Count of Participants; unit: Participants]
  Participants with 1 Previous Line of Chemotherapy | 0
  Participants with 2 Previous Lines of Chemotherapy | 2
  Participants with 3 Previous Lines of Chemotherapy | 5
  Participants with 4 Previous Lines of Chemotherapy | 5
  Participants with 5 Previous Lines of Chemotherapy | 5
  Participants with 6 Previous Lines of Chemotherapy | 1

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Serious Adverse Events Rate
Description: Freedom from Serious Adverse Events reports the number of participants that did not have a serious adverse event reported within 30 days of treatment that results in any of the following outcomes: Death, a life-threatening adverse drug experience, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defects.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 40um Embozene TANDEM Microspheres
Number analyzed (Participants) | 18
Participants | 18

2. Primary Outcome: Local Tumor Control
Description: Local tumor control reports the percent of subjects for which the size of the tumor does not increase. Local Tumor Control is defined as subjects having complete response or stable disease. For these subjects the treated tumor either shrinks or stays the same size when measuring the tumor using a standard tumor measurement guideline (based on the devascularization pattern from the European Association for the Study of the Liver (EASL) criteria).
Time Frame: 3 months post procedure
Population: All subjects were included in this analysis except for one subject that was removed from the study after undergoing liver resection surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | 40um Embozene TANDEM Microspheres
Number analyzed (Participants) | 17
Participants | 15

3. Primary Outcome: Local Tumor Control
Description: as for outcome 2
Time Frame: 6 months post procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 40um Embozene TANDEM Microspheres
Number analyzed (Participants) | 17
Participants | 7

4. Primary Outcome: Local Tumor Control
Description: as for outcome 2
Time Frame: 12 months post procedure
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 40um Embozene TANDEM Microspheres
Number analyzed (Participants) | 17
Participants | 3

5. Secondary Outcome: Survival Rate
Description: Number of participants that were alive 12 months after their first study treatment.
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | 40um Embozene TANDEM Microspheres
Number analyzed (Participants) | 18
Participants | 10

6. Secondary Outcome: Time To Tumor Progression
Description: Time to Tumor Progression is defined as the time from the date of first study treatment to the day of documented disease progression or death due to any cause, whichever came first, assessed up to 1 year. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (mRECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 12 months post procedure
Population: Two participants that did not have disease progression reported during the trial are not included in this analysis. One subject underwent liver resection surgery after their third study treatment and another subject's tumor response was reported as stable disease prior to being lost to follow up after their third study treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 40um Embozene TANDEM Microspheres
Number analyzed (Participants) | 16
days | 177.2 (111.4)

ADVERSE EVENTS:
Time Frame: Up to 24 months post procedure
Arm/Group | 40um Embozene TANDEM Microspheres
All-Cause Mortality (participants affected / at risk) | 10/18
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40um Embozene TANDEM Microspheres (N=18)
Progression of Disease (Hepatobiliary disorders) | 10 (10) — Progression of Disease leading to death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40um Embozene TANDEM Microspheres (N=18)
Post Embolization Syndrome (General disorders) | 14 (28) — Abdominal Pain, Nausea, Fatigue & Fever
Decreased Liver Function (Hepatobiliary disorders) | 6 (8) — Total Bilirubin Increase
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Allergic Reaction (Immune system disorders) | 2 (2) — Allergic Reaction to Contrast Media
Asthenia (General disorders) | 1 (1) — Abnormal physical weakness or lack of energy
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Anorexia (General disorders) | 1 (1)
Bone Fracture (Injury, poisoning and procedural complications) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) — The presence of abnormally few neutrophils in the blood, leading to increased susceptibility to infection
Edema (General disorders) | 1 (1) — A condition characterized by an excess of watery fluid collecting in the cavities or tissues of the body.
Access Site Haemorrhage (Surgical and medical procedures) | 1 (1)
Hypochondrium Pain (General disorders) | 1 (2) — Abdominal pain
Visual Impairment (Eye disorders) | 1 (1) — Accommodation Disorder

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No